CLINICAL TRIAL: NCT07096674
Title: A Phase 2, Long-term Extension Study of the Safety and Efficacy of ORX750 in Participants With Narcolepsy and Idiopathic Hypersomnia Who Completed a Sponsored ORX750 Clinical Trial
Brief Title: A Long-term Extension Study of ORX750 in Participants With Narcolepsy and Idiopathic Hypersomnia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centessa Pharmaceuticals (UK) Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORX750-202
Record Dates: First submitted 2025-07-02; First posted 2025-07-31 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Narcolepsy Type 1; Narcolepsy Type 2; Idiopathic Hypersomnia
Keywords: NT1; NT2; IH; Narcolepsy; Narcolepsy Type 1; Narcolepsy Type 2; Idiopathic Hypersomnia; Excessive Daytime Sleepiness; Orexin Receptor 2 agonist
MeSH Terms: conditions — Idiopathic Hypersomnia; Narcolepsy; Disorders of Excessive Somnolence

STUDY DESIGN:
Intervention Model Description: Open Label Long Term Extension Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Narcolepsy Type 1 (Experimental): Narcolepsy Type 1 (Open Label)
  Interventions: Drug: ORX750
- Narcolepsy Type 2 (Experimental): Narcolepsy Type 2 (Open Label)
  Interventions: Drug: ORX750
- Idiopathic Hypersomnia (Experimental): Idiopathic Hypersomnia (Open Label)
  Interventions: Drug: ORX750

INTERVENTIONS:
Drug: ORX750 — Oral ORX750
  Arms: Narcolepsy Type 1
Drug: ORX750 — Oral ORX750
  Arms: Narcolepsy Type 2
Drug: ORX750 — Oral ORX750
  Arms: Idiopathic Hypersomnia

SUMMARY:
This study is a long-term extension (LTE) of the parent Study ORX750 0201, and will provide long-term open-label safety, tolerability, and efficacy of ORX750 in participants with narcolepsy type 1 (NT1), narcolepsy type 2 (NT2), and idiopathic hypersomnia (IH).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of narcolepsy (NT1 or NT2) or IH who was eligible for and completed the full treatment period in the eligible parent study ORX750-0201 (CRYSTAL-1)
* Is willing and able to adhere to additional protocol requirements

Exclusion Criteria:

* Development of any new disease/disorder that in the opinion of the investigator would make the participant unable to continue the study
* Unable to refrain from excluded medications, including those used for treatment of narcolepsy or idiopathic hypersomnia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs | Up to day 70
  Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Abnormal Laboratory Tests | Up to day 70
  Number of Participants With Abnormal Changes From Baseline in Laboratory Tests
Abnormal Vital Signs | Up to day 70
  Number of Participants With Abnormal Change From Baseline in Vital Signs
Abnormal ECG | Up to day 70
  Number of Participants With Abnormal Change From Baseline in Electrocardiograms (ECG)
Suicidal Ideation or Behavior | Up to day 70
  Number of Participants With Suicidal Ideation or Suicidal Behavior as Measured Using Columbia-Suicide Severity Rating Scale (C-SSRS)

SECONDARY OUTCOMES:
Cmax | Up to day 63
  Cmax: Maximum Observed Plasma Concentration for ORX750
Tmax | Up to day 63
  Tmax: Time of Maximum Concentration for ORX750
AUClast | Up to day 63
  AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for ORX750
Cmax,ss | Up to day 63
  Cmax,ss: Maximum Observed Concentration at Steady State for ORX750
AUCτ | Up to day 63
  AUCτ: Area Under the Concentration-time Curve During a Dosing Interval at Steady State for ORX750
Maintenance of Wakefulness Test | Up to day 63
  Change From Baseline in Mean sleep latency (average of the first 4 trials) in the Maintenance of Wakefulness Test (MWT)
Epworth Sleepiness Scale | Up to day 63
  Change From Baseline in Epworth Sleepiness Scale (ESS)

CONTACTS AND LOCATIONS:
Locations (1):
- Site Number 1, Huntersville, North Carolina, United States